CLINICAL TRIAL: NCT02112136
Title: Clinical and Molecular Description of PKD1 and PKD2 Mutation Negative Carriers in Autosomal Dominant Polycystic Kidney Disease (ADPKD): The GeneQuest Study
Brief Title: Clinical and Molecular Description of PKD1 and PKD2 Mutation Negative Carriers in ADPKD
Acronym: GeneQuest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RB14.017 GeneQuest
Record Dates: First submitted 2014-04-09; First posted 2014-04-11 (Estimated); Last update posted 2021-03-24 (Actual); Status verified 2020-12

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Keywords: Autosomal Dominant Polycystic Kidney Disease (ADPKD); Renal cysts; Chronic Kidney Diseases; Genetic
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Renal Insufficiency, Chronic | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GeneQuest (Other): * No drug will be administrated in this study
  * Blood collection
  Interventions: Other: Blood Collection

INTERVENTIONS:
Other: Blood Collection — Phenotype and Genotype Analysis, Biological Analysis

SUMMARY:
The aim of this study is to identify families with ADPKD , characterize the phenotype and screen for mutations in known genes (PKD1 and PKD2, and then HNF1b and UMOD in PKD1 PKD2 negative carriers).

Genome wide analysis will be performed in families without mutations identified.

DETAILED DESCRIPTION:
* Inclusion of ADPKD patients in 20 different centers of Nephrology in the Western part of France
* Characterization of the Phenotype
* Collect DNA sample
* Analysis of PKD1 and PKD2 genes first
* Analysis of HNFIb and UMOD for PKD1 and PKD2 negative patients
* Recruitment of affected and non-affected relatives of PKD1 and PKD2 negative ADPKD patients
* Identify new genes involved in ADPKD using exome sequencing in PKD1 and PKD2 negative pedigrees

ELIGIBILITY:
Inclusion Criteria for the proband :

* Patients with a diagnosis of ADPKD
* Written Informed Consent
* Affiliated or benefiting from a national insurance

Inclusion Criteria of the relatives (affected or non affected) :

* Relatives with a diagnosis of ADPKD (ADPKD relatives)
* And Relatives over age 30 for whom the diagnosis of ADPKD has been discarded (non ADPKD relatives) with renal ultrasonography performed after age 30.
* Written Informed consent
* Affiliated or benefiting from a national insurance

Exclusion Criteria for the Probands:

* Subjects unable to provide written informed consent
* Previous Molecular analysis of PKD1 and PKD2 genes with identification of the pathogenic mutation

Exclusion criteria for the Relatives:

* Subjects unable to provide written informed consent
* Age under 30 for the "non-affected" relatives

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1450 (Actual)
Dates: Start 2014-12-12 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
Number of patients/families with no mutations identified in PKD1 and PKD2 genes | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Cornec-Le Gall, MD, Principal Investigator — CHRU de Brest
Locations (25):
- France (25):
  - CHU Angers, Angers
  - AUB Brest, Brest
  - Centre de néphrologie et de dialyse d'Armorique, Brest
  - CHRU Brest, Brest
  - CH Laval, Laval
  - CH du Mans, Le Mans
  - ECHO dialyse, Le Mans
  - Centre de dialyse de Lorient, Lorient
  - CH Bretagne Sud, Lorient
  - Hôpital Hôtel Dieu - CHU Nantes, Nantes
  - CH Niort, Niort
  - ECHO les Sables d'Olonne, Olonne-sur-Mer
  - Hôpital Jean Bernard - CHU Poitiers, Poitiers
  - CHCB site de Noyal Pontivy, Pontivy
  - CH Laënnec, Quimper
  - AUB Santé, Quimper
  - Hôpital Pontchaillou, Rennes
  - Echo Csmn, Rezé
  - Centre de Pérharidy, Roscoff
  - Hôpital Yves Le Foll, Saint-Brieuc
  - ECHO Centre Ambulatoire, Saint-Herblain
  - CH de Saint Nazaire, Saint-Nazaire
  - CH Saint Malo, St-Malo
  - Hôpital Bretonneau - CHU Tours, Tours
  - CH Bretagne Atlantique - Site de Vannes, Vannes

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning one year and ending fifteen years following the final study report completion
Access Criteria: Data access will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement

REFERENCES:
- [Derived] Lefevre S, Audrezet MP, Halimi JM, Longuet H, Bridoux F, Ecotiere L, Augusto JF, Duveau A, Renaudineau E, Vigneau C, Frouget T, Charasse C, Gueguen L, Perrichot R, Couvrat G, Seret G, Le Meur Y, Cornec-Le Gall E; Genkyst Study Group. Diagnosis and risk factors for intracranial aneurysms in autosomal polycystic kidney disease: a cross-sectional study from the Genkyst cohort. Nephrol Dial Transplant. 2022 Oct 19;37(11):2223-2233. doi: 10.1093/ndt/gfac027. PMID 35108395